CLINICAL TRIAL: NCT04748146
Title: CAUSAL MECHANISMS OF DISTRIBUTED BRAIN NETWORK FUNCTION DURING EPISODIC MEMORY RETRIEVAL
Brief Title: In-depth Investigation of Brain Network Interactions
Acronym: BNI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was withdrawn due to changes in the study design or protocol.
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU00213066
Record Dates: First submitted 2021-02-08; First posted 2021-02-10 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Episodic Memory
Keywords: Episodic Memory; Default Network; Brain Stimulation
MeSH Terms: interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: All participants will receive theta-burst stimulation and sham stimulation, meaning that each participant will be their own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention and Control group (Other): Each patient will receive electrical and sham stimulation, meaning that each patient will act as their own control.
  Interventions: Other: Brain stimulation

INTERVENTIONS:
Other: Brain stimulation — Theta-burst stimulation will be applied to selected regions of distributed networks to test whether distal stimulation can modulate hippocampus-mediated episodic recollection.

SUMMARY:
Brain stimulation is a means to potentially remediate symptoms in a range of neurological and psychiatric diseases, however, precise targeting of stimulation is necessary to ensure efficacy. The proposed project will use recent advances in functional magnetic resonance imaging to delineate distributed brain networks within individuals, and use these network maps to guide selection of intracranial electrodes for stimulation during an episodic memory task. The resulting data will refine the current understanding of the neural systems involved in episodic memory, and provide a proof-of-principle for the use of individual-level network mapping to guide brain stimulation, which could have important implications for brain stimulation therapies for a range of mental health disorders.

DETAILED DESCRIPTION:
Research Statement SIGNIFICANCE Memory impairments are common to several neurological and psychiatric disorders, including Alzheimer's disease and depression, and these impose a heavy burden on patients, families and society (Dickerson and Eichenbaum, 2007). Novel treatment and diagnostic strategies are needed, and these may arise from a deeper understanding of the brain basis of episodic memory (Tulving, 1983).

Group-averaged neuroimaging studies have revealed that a distributed network, known as the 'default network' (DN), increases activity during the recollection of past events (Buckner et al. 2008). This network occupies regions including posteromedial cortex (PMC), posterior parietal cortex (PPC), and the medial temporal lobe (MTL), as well as lateral temporal and lateral and medial prefrontal cortices. Building on recent advances in functional magnetic resonance imaging (fMRI; Poldrack et al., 2015; Laumann et al., 2015), recent evidence has shown that when functional anatomy is defined in individuals, the DN comprises at least two juxtaposed networks, named DN-A and DN-B for convenience (Figure 1). This finding forces us to reconsider the role of the DN in episodic processes (see also: Dastjerdi et al., 2011; Andrews-Hanna et al., 2010). Here we propose experiments to deepen our understanding of these networks using a multimodal approach that provides high spatiotemporal resolution and whole-brain network definition. We will combine within-individual fMRI mapping with intracranial electroencephalography (iEEG) and electrical brain stimulation (EBS). We will directly record local field potentials from precisely mapped network regions, and apply electrical stimulation with millimeter precision. This will provide novel information regarding episodic memory in two domains that cannot be gathered by fMRI alone: i) characterizing fast temporal dynamics of network recruitment during episodic recollection, and ii) establishing causal interactions between brain regions during recollection.

INNOVATION Methodologically, this project will provide proof of principle that precision fMRI mapping can be performed in a clinical population and successfully combined with invasive recordings and stimulation. Theoretical innovation will be obtained through a deeper understanding of the task-response dynamics, coupling, and causal relationships between regions of distributed networks, including how neural engagement changes during memory recollection. Finally, this proposal provides translational innovation by directly testing whether precision-fMRI guided intracranial stimulation can be used modulate memory performance.

APPROACH General methods: Participants in the proposed experiments will be neurosurgical patients with presumed focal epilepsy that are to undergo implantation with intracranial electrodes for localizing seizure foci. The proposal will be carried out at the Northwestern University Feinberg School of Medicine. Patients scheduled for intracranial seizure monitoring will be invited to enroll in the study and will undergo 1 to 4 sessions of fMRI prior to surgical implantation of electrodes. After surgery, patients are typically monitored for ~7 days in the Northwestern Memorial Hospital Comprehensive Epilepsy Centre (CEC), during which they will be invited to participate in the proposed experiments. All subjects must provide informed consent before participating.

Enrollment: A minimum of 40-50 patients are expected to be monitored at the CEC over the next 3 years. Electrode locations are determined by the clinical needs of the patient. 60-70% of patients are typically implanted with dense coverage of the medial temporal lobes achieved through depth electrodes with trajectories that allow sampling of lateral temporal cortices. A small number of electrodes are also typically implanted in posterior cingulate, lateral inferior parietal and ventromedial prefrontal cortex. Due to the distributed nature of the networks under investigation, which contain regions in multiple cortical zones, it is likely that we will have coverage over relevant brain regions in many cases. Some patients are also likely to be implanted with broader cortical coverage using subdural grids. Preliminary results have shown that even when a patient is implanted only with depth electrodes, which are not placed on the cortical surface but penetrate into the brain, coverage of different candidate network regions was often achieved along the electrode trajectory. With conservative estimates, 20-30 subjects will be good candidates for the project aims outlined below. Given the high signal-to-noise ratio of iEEG (usually a 200-300% task-evoked increase in signal from baseline; Parvizi and Kastner, 2017), reliable effects can typically be found within individuals. All proposed analyses will be carried out within individuals, hence multiple subjects are required to generalize the findings, not increase statistical power. Therefore, a small number of subjects (as low as n = 12) would be sufficient (e.g. Braga and Buckner, 2017; Foster et al., 2013).

Neuroimaging acquisition: MR scans will be collected in 1-4 sessions from each patient. Preliminary data has shown that in this clinical population 2-3 MRI sessions are desirable to allow exclusion of non-compliant runs (e.g. those containing excess head motion). We will collect 6-8 runs of fMRI data per session, resulting in between 42 - 224 mins of fMRI data per patient. This will allow robust and reliable estimates of network topography. Subject sleepiness will be monitored through an in-scanner eye-tracking camera. Compliance may be improved by allowing patients to watch movies inside the scanner when needed, with pilot analyses showing comparable maps are obtained using movie and visual fixation task data. Hence both tasks will be administered to improve compliance.

Network definition within individuals: Networks will be defined within individuals using two methods to ensure robustness. MRI preprocessing will be performed using a custom pipeline 'iProc' that optimizes within-subject alignment and minimizes blurring. Individual seed regions will be hand-selected and correlation maps will be thresholded at r > 0.2 to remove regions of low certainty. The networks of interest, DN-A and DN-B, will be targeted and identified using the expected anatomical distribution of each network (described in detail in Braga and Buckner, 2017). Once candidate seed regions are selected, definition of networks will be performed again in each individual using data-driven clustering, which reduces potential experimenter bias. Networks from the clustering analysis that most closely match up with the networks defined by hand will be selected and labelled as DN-A and DN-B. Network maps will be used to label electrode contacts (each 'electrode' can have multiple 'contacts' along its shaft or grid) by their approximate location within or near each network.

Electrode localization: Electrode locations will be determined using a computerized tomography (CT) scan. Estimates of the center of each contact in CT space will be obtained using BioImage Suite. The CT image will be registered to the anatomical T1 image (containing brain tissue locations) using a linear transform, allowing coordinates of each contact to be projected to the T1 space. Preliminary data has shown that the inter-rater error in this localization process is typically ~1mm. A 2-mm radius sphere will be generated centered on each contact coordinate to approximate the sampling volume of each contact, which is extended due to tissue conductance. Contacts that are predominantly sampling white matter will be removed by excluding contacts whose sphere does not overlap with the gray matter ribbon (estimated using FreeSurfer). The overlap between spheres and gray matter will be used for surface-based and volume-based functional connectivity (FC) analyses. FC maps will be created for each contact, and the resulting maps will be visualized. If a contact fails to produce a FC map with distant regions of high correlation (indicating that the contact is sampling a distributed network), the contact will be excluded. If the contact's FC map resembles DN-A and DN-B, as defined using the clustering and manually defined seed-based analyses, this contact will be labelled as sampling DN-A and DN-B and included for further analysis. Two nearby electrodes, one situated in DN-A and one in DN-B, will be selected a priori in two different cortical zones (e.g. PMC vs. PPC, based on coverage).

iEEG processing: All contacts within the epileptic zone or corrupted by external noise will be removed from further analysis. Raw signals will be notch filtered at 60, 120 and 180 Hz to remove electrical noise and harmonics. Notch-filtered signals will be re-referenced by subtracting the common average, after removal of pathogenic or spiky signals, as well as those presenting as clear outliers in power spectra plots. Data will be bandpass filtered to extract amplitude and phase information at different frequency bands. The high-frequency broadband (HFB; 70-140 Hz) signal is an important surrogate for local neuronal population activity and corresponds to low-frequency correlations of the blood oxygenation-level dependent signal (Logothetis et al., 2001). HFB band-limited power will be calculated and low-pass filtered at <0.1 Hz. Pair-wise correlations in HFB power will be used to estimate functional connectivity.

Direct cortical stimulation: Risks associated with the research stimulation protocol are considered incremental and are further reduced by carrying out the stimulation under supervision of a clinical researcher, when patients are on antiepileptic medication, and keeping stimulation to within safety limits. Low frequency (1 Hz) single pulse stimulation will be applied to regions of DN-A and DN-B to map cortico-cortical evoked potentials (CCEPs). This will be used to estimate the strength, as well as provide data on the directionality of connections between regions. In a departure from original plans, based on recent findings (Hermiller et al. 2019), theta-burst stimulation (gamma-band stimulation applied intermittently at theta frequencies) will be applied to regions of DN-A regions in lateral temporal, posteromedial and prefrontal cortices during a recollection task to test if stimulation of distant DN-A regions can lead to improvements in hippocampus-mediated episodic memory recollection. Currents will be administered at a threshold below that which causes after-discharges (usually around 6-8 mA).

ELIGIBILITY:
Participants will be inpatients of the Northwestern Memorial Hospital Comprehensive Epilepsy Center undergoing intracranial electroencephalography for presurgical planning as part of their routine care for epilepsy. Participants will be recruited to participate in the study if their epilepsy monitoring procedures will include placement of recording electrodes at locations of interest to our study, which include the medial temporal lobe, frontal cortex, parietal cortex, and temporal cortex. The decision regarding where to place electrodes is made for purely clinical purposes and we recruit patients with locations that are relevant to our research question as a convenience sample.

We will exclude children under the age of 18 years as brain development is still occurring in children under the age of 18 years relative to adults. Furthermore, children rarely receive iEEG for epilepsy and therefore would not be available to recruit into the study. Special populations listed below will not participate in this study. Excluded populations include:

1. Adults legally unable to provide informed consent
2. Individuals who are not yet adults (children below the age of 18)
3. Pregnant women
4. Prisoners To help determine eligibility for the MRI portion of the study, a safety questionnaire will be administered by research staff prior to receiving an MRI. Answers to these questions are used to determine whether subjects meet any of the exclusionary criteria listed next. Exclusions for MRI include standard MRI contraindications, including claustrophobia, metal implants or fragments in the body, and actual or potential pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Reaction Time | Immediate during procedure
  Reaction time for cued episodic recollection task
Accuracy | Immediate during procedure
  Number of correct responses in cued episodic recollection task

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo M Braga, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tulving, E. (1983) Elements of episodic memory. Oxford. Clarendon Press ; New York : Oxford University Press. xi, 351 p. p.
- [Background] Dickerson BC, Eichenbaum H. The episodic memory system: neurocircuitry and disorders. Neuropsychopharmacology. 2010 Jan;35(1):86-104. doi: 10.1038/npp.2009.126. PMID 19776728
- [Background] Buckner RL, Andrews-Hanna JR, Schacter DL. The brain's default network: anatomy, function, and relevance to disease. Ann N Y Acad Sci. 2008 Mar;1124:1-38. doi: 10.1196/annals.1440.011. PMID 18400922
- [Background] Poldrack RA, Laumann TO, Koyejo O, Gregory B, Hover A, Chen MY, Gorgolewski KJ, Luci J, Joo SJ, Boyd RL, Hunicke-Smith S, Simpson ZB, Caven T, Sochat V, Shine JM, Gordon E, Snyder AZ, Adeyemo B, Petersen SE, Glahn DC, Reese Mckay D, Curran JE, Goring HH, Carless MA, Blangero J, Dougherty R, Leemans A, Handwerker DA, Frick L, Marcotte EM, Mumford JA. Long-term neural and physiological phenotyping of a single human. Nat Commun. 2015 Dec 9;6:8885. doi: 10.1038/ncomms9885. PMID 26648521
- [Background] Laumann TO, Gordon EM, Adeyemo B, Snyder AZ, Joo SJ, Chen MY, Gilmore AW, McDermott KB, Nelson SM, Dosenbach NU, Schlaggar BL, Mumford JA, Poldrack RA, Petersen SE. Functional System and Areal Organization of a Highly Sampled Individual Human Brain. Neuron. 2015 Aug 5;87(3):657-70. doi: 10.1016/j.neuron.2015.06.037. Epub 2015 Jul 23. PMID 26212711
- [Background] Andrews-Hanna JR, Reidler JS, Sepulcre J, Poulin R, Buckner RL. Functional-anatomic fractionation of the brain's default network. Neuron. 2010 Feb 25;65(4):550-62. doi: 10.1016/j.neuron.2010.02.005. PMID 20188659
- [Background] Braga RM, Buckner RL. Parallel Interdigitated Distributed Networks within the Individual Estimated by Intrinsic Functional Connectivity. Neuron. 2017 Jul 19;95(2):457-471.e5. doi: 10.1016/j.neuron.2017.06.038. PMID 28728026
- [Background] Dastjerdi M, Foster BL, Nasrullah S, Rauschecker AM, Dougherty RF, Townsend JD, Chang C, Greicius MD, Menon V, Kennedy DP, Parvizi J. Differential electrophysiological response during rest, self-referential, and non-self-referential tasks in human posteromedial cortex. Proc Natl Acad Sci U S A. 2011 Feb 15;108(7):3023-8. doi: 10.1073/pnas.1017098108. Epub 2011 Jan 31. PMID 21282630
- [Background] DiNicola LM, Braga RM, Buckner RL. Parallel distributed networks dissociate episodic and social functions within the individual. J Neurophysiol. 2020 Mar 1;123(3):1144-1179. doi: 10.1152/jn.00529.2019. Epub 2020 Feb 12. PMID 32049593
- [Background] Foster BL, Kaveh A, Dastjerdi M, Miller KJ, Parvizi J. Human retrosplenial cortex displays transient theta phase locking with medial temporal cortex prior to activation during autobiographical memory retrieval. J Neurosci. 2013 Jun 19;33(25):10439-46. doi: 10.1523/JNEUROSCI.0513-13.2013. PMID 23785155
- [Background] Foster BL, Parvizi J. Direct cortical stimulation of human posteromedial cortex. Neurology. 2017 Feb 14;88(7):685-691. doi: 10.1212/WNL.0000000000003607. Epub 2017 Jan 18. PMID 28100728
- [Background] Hebscher M, Voss JL. Testing network properties of episodic memory using non-invasive brain stimulation. Curr Opin Behav Sci. 2020 Apr;32:35-42. doi: 10.1016/j.cobeha.2020.01.012. Epub 2020 Feb 28. PMID 32266318
- [Background] Hermiller MS, VanHaerents S, Raij T, Voss JL. Frequency-specific noninvasive modulation of memory retrieval and its relationship with hippocampal network connectivity. Hippocampus. 2019 Jul;29(7):595-609. doi: 10.1002/hipo.23054. Epub 2018 Dec 11. PMID 30447076
- [Background] Logothetis NK, Pauls J, Augath M, Trinath T, Oeltermann A. Neurophysiological investigation of the basis of the fMRI signal. Nature. 2001 Jul 12;412(6843):150-7. doi: 10.1038/35084005. PMID 11449264
- [Background] Parvizi J, Kastner S. Promises and limitations of human intracranial electroencephalography. Nat Neurosci. 2018 Apr;21(4):474-483. doi: 10.1038/s41593-018-0108-2. Epub 2018 Mar 5. PMID 29507407
- [Background] Suthana N, Haneef Z, Stern J, Mukamel R, Behnke E, Knowlton B, Fried I. Memory enhancement and deep-brain stimulation of the entorhinal area. N Engl J Med. 2012 Feb 9;366(6):502-10. doi: 10.1056/NEJMoa1107212. PMID 22316444
- [Background] Wang L, Saalmann YB, Pinsk MA, Arcaro MJ, Kastner S. Electrophysiological low-frequency coherence and cross-frequency coupling contribute to BOLD connectivity. Neuron. 2012 Dec 6;76(5):1010-20. doi: 10.1016/j.neuron.2012.09.033. PMID 23217748